CLINICAL TRIAL: NCT06743516
Title: The Impact of External Pancreatic Drainage During Pancreaticojejunostomy Following Pancreaticoduodenectomy in Cases of Soft Pancreas
Brief Title: External Pancreatic Stent in Pancreaticojejunostomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Saleh Khairy Saleh MD, Lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1282/10/2024
Record Dates: First submitted 2024-12-12; First posted 2024-12-20 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Fistula
MeSH Terms: conditions — Pancreatic Fistula | interventions — Pancreaticojejunostomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Surgeons are not blinded due to the intervention's nature; data collectors, assessors, and analysts are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pancreaticojejunostomy with External stent (Active Comparator): ureteric catheter (7Fr) insert at pancreatojejunostomy site as a stent. And stent tube is brought out through jejunal loop below the hepaticojejunostomy site and abdominal wall.
  Interventions: Procedure: Pancreaticojejunostomy with external stent
- Pancreaticojejunostomy without stent (Active Comparator): Pancreaticojejunostomy without stent
  Interventions: Procedure: Pancreaticojejunostomy without external stent

INTERVENTIONS:
Procedure: Pancreaticojejunostomy with external stent — Inserting ureteric stent at the pancreaticojejunostomy site
  Arms: Pancreaticojejunostomy with External stent
Procedure: Pancreaticojejunostomy without external stent — Only Pancreaticojejunostomy without inserting external stent
  Arms: Pancreaticojejunostomy without stent

SUMMARY:
Pancreatic fistula is one of the most serious complication after pancreatoduodenectomy. To reduce pancreatic fistula, many authors recommend pancreatic stent in pancreatojejunostomy. The purpose of this study is to determine which is the best method in preventing pancreatic fistula and to investigate its long term clinical outcomes.

DETAILED DESCRIPTION:
The role of external pancreatic duct drainage in managing patients with a soft pancreas is particularly important, as these patients are at a heightened risk of developing postoperative complications. By providing an external route for pancreatic secretions, external pancreatic duct drainage may help to reduce the enzymatic activity at the anastomosis site and promote better healing.

In addition to reducing the incidence of post operative pancreatic fistula, external pancreatic duct drainage may have other potential benefits, such as decreasing the length of hospital stay, reducing the need for additional interventions, and improving overall patient quality of life. However, these potential benefits must be weighed against the risks and drawbacks of external pancreatic duct drainage, including the potential for stent-related complications and the need for an additional procedure to remove the stent.

•After being informed about the study and potential risks, all patients giving written consent. Patients who meet the eligibility requirements will be randomized in a 1:1 ratio to external pancreatic drainage group and no external pancreatic drainage group.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pancreaticoduodenectomy (Whipple procedure) for various indications (e.g., pancreatic cancer, ampullary cancer, etc.).
* Patients with a confirmed soft pancreas texture, as determined intraoperatively by the surgeon.

Exclusion Criteria:

* Patients with a hard or fibrotic pancreas, as determined intraoperatively by the surgeon.
* Patients with severe uncontrolled comorbidities (e.g., uncontrolled diabetes, severe cardiovascular disease, renal failure).
* Pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
evidence of pancreatic fistula | within the first 7 days after surgery( first day, third day and fifth day)
  confirmed by serum and drain amylase

SECONDARY OUTCOMES:
evidence of intra abdominal collection | first week, second week postoperative
  confirmed by abdominal ultrasound and abdominal computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Saleh K Saleh, MD, Principal Investigator — Minia University
Locations (1):
- Liver and GIT hospital , Minia University, Minya, Egypt